CLINICAL TRIAL: NCT01379339
Title: Phase I Study of Cabazitaxel - Platinum Fluorouracil Induction Chemotherapy in Patients With Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Cabazitaxel - PF Induction Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Krzysztof Misiukiewicz (Other)
Collaborators: Sanofi (Industry); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor-Investigator, Krzysztof Misiukiewicz, Assistant Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 11-0646(0001)(01); 183133-96-2 (Registry Identifier: CAS Registry); HS#: 11-00201
Record Dates: First submitted 2011-06-15; First posted 2011-06-23 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Cabazitaxel; Cabazitaxel and Cisplatin; Phase I; PF Induction Chemotherapy; Squamous Cell Carcinoma; Head and Neck; Sanofi-Aventis Oncology; Locally Advanced
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell | interventions — cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cabazitaxel 10mg/m2 (Experimental): * Cabazitaxel on D1 Dose: 10mg/m2 IV x 1 Route: Intravenous infusion over 60 minutes, mixed as described in protocol over 1 hour Schedule: Day 1, every 21 days (+ 2 days)
  * Cisplatin on D1 Dose: 100 mg/m2 Route: Intravenous infusion over 60 minutes to 3 hours, mixed in 1000 ml of normal saline Schedule: Day 1, every 21 days (+ 2 days)
  * 5 Fluorouracil on D1-D4 Dose: 800 mg/m2/day Route: 24-hour continuous infusion over 4 days Schedule: Days 1, 2, 3 and 4 of Cycles 1, 2 and 3 (every 21 days) + 2 days)
  Interventions: Drug: Cabazitaxel 10mg/m2
- Cabazitaxel 12.5mg/m2 (Experimental): * Cabazitaxel on D1 Dose: 12.5mg/m2 IV x 1 Route: Intravenous infusion over 60 minutes, mixed as described in protocol over 1 hour Schedule: Day 1, every 21 days (+ 2 days)
  * Cisplatin on D1 Dose: 100 mg/m2 Route: Intravenous infusion over 60 minutes to 3 hours, mixed in 1000 ml of normal saline Schedule: Day 1, every 21 days (+ 2 days)
  * 5 Fluorouracil on D1-D4 Dose: 800 mg/m2/day Route: 24-hour continuous infusion over 4 days Schedule: Days 1, 2, 3 and 4 of Cycles 1, 2 and 3 (every 21 days) + 2 days)
  Interventions: Drug: Cabazitaxel 12.5mg/m2
- Cabazitaxel 15mg/m2 (Experimental): * Cabazitaxel on D1 Dose: 15mg/m2 IV x 1 Route: Intravenous infusion over 60 minutes, mixed as described in protocol over 1 hour Schedule: Day 1, every 21 days (+ 2 days)
  * Cisplatin on D1 Dose: 100 mg/m2 Route: Intravenous infusion over 60 minutes to 3 hours, mixed in 1000 ml of normal saline Schedule: Day 1, every 21 days (+ 2 days)
  * 5 Fluorouracil on D1-D4 Dose: 800 mg/m2/day Route: 24-hour continuous infusion over 4 days Schedule: Days 1, 2, 3 and 4 of Cycles 1, 2 and 3 (every 21 days) + 2 days)
  Interventions: Drug: Cabazitaxel 15mg/m2
- Cabazitaxel 17.5mg/m2 (Experimental): * Cabazitaxel on D1 Dose: 17.5mg/m2 IV x 1 Route: Intravenous infusion over 60 minutes, mixed as described in protocol over 1 hour Schedule: Day 1, every 21 days (+ 2 days)
  * Cisplatin on D1 Dose: 100 mg/m2 Route: Intravenous infusion over 60 minutes to 3 hours, mixed in 1000 ml of normal saline Schedule: Day 1, every 21 days (+ 2 days)
  * 5 Fluorouracil on D1-D4 Dose: 800 mg/m2/day Route: 24-hour continuous infusion over 4 days Schedule: Days 1, 2, 3 and 4 of Cycles 1, 2 and 3 (every 21 days) + 2 days)
  Interventions: Drug: Cabazitaxel 17.5mg/m2
- Cabazitaxel 20mg/m2 (Experimental): * Cabazitaxel on D1 Dose: 20mg/m2 IV x 1 Route: Intravenous infusion over 60 minutes, mixed as described in protocol over 1 hour Schedule: Day 1, every 21 days (+ 2 days)
  * Cisplatin on D1 Dose: 100 mg/m2 Route: Intravenous infusion over 60 minutes to 3 hours, mixed in 1000 ml of normal saline Schedule: Day 1, every 21 days (+ 2 days)
  * 5 Fluorouracil on D1-D4 Dose: 800 mg/m2/day Route: 24-hour continuous infusion over 4 days Schedule: Days 1, 2, 3 and 4 of Cycles 1, 2 and 3 (every 21 days) + 2 days)
  Interventions: Drug: Cabazitaxel 20mg/m2

INTERVENTIONS:
Drug: Cabazitaxel 10mg/m2 — * Cabazitaxel on D1 Dose: 10mg/m2 IV x 1 Route: Intravenous infusion over 60 minutes, mixed as described in protocol over 1 hour Schedule: Day 1, every 21 days (+ 2 days)
  * Cisplatin on D1 Dose: 100 mg/m2 Route: Intravenous infusion over 60 minutes to 3 hours, mixed in 1000 ml of normal saline Schedule: Day 1, every 21 days (+ 2 days)
  * 5 Fluorouracil on D1-D4 Dose: 800 mg/m2/day Route: 24-hour continuous infusion over 4 days Schedule: Days 1, 2, 3 and 4 of Cycles 1, 2 and 3 (every 21 days) + 2 days)
  Other Names: Cabazitaxel-PF Induction Chemotherapy
  Arms: Cabazitaxel 10mg/m2
Drug: Cabazitaxel 12.5mg/m2 — * Cabazitaxel on D1 Dose: 12.5mg/m2 IV x 1 Route: Intravenous infusion over 60 minutes, mixed as described in protocol over 1 hour Schedule: Day 1, every 21 days (+ 2 days)
  * Cisplatin on D1 Dose: 100 mg/m2 Route: Intravenous infusion over 60 minutes to 3 hours, mixed in 1000 ml of normal saline Schedule: Day 1, every 21 days (+ 2 days)
  * 5 Fluorouracil on D1-D4 Dose: 800 mg/m2/day Route: 24-hour continuous infusion over 4 days Schedule: Days 1, 2, 3 and 4 of Cycles 1, 2 and 3 (every 21 days) + 2 days)
  Other Names: Cabazitaxel-PF Induction Chemotherapy
  Arms: Cabazitaxel 12.5mg/m2
Drug: Cabazitaxel 15mg/m2 — * Cabazitaxel on D1 Dose: 15mg/m2 IV x 1 Route: Intravenous infusion over 60 minutes, mixed as described in protocol over 1 hour Schedule: Day 1, every 21 days (+ 2 days)
  * Cisplatin on D1 Dose: 100 mg/m2 Route: Intravenous infusion over 60 minutes to 3 hours, mixed in 1000 ml of normal saline Schedule: Day 1, every 21 days (+ 2 days)
  * 5 Fluorouracil on D1-D4 Dose: 800 mg/m2/day Route: 24-hour continuous infusion over 4 days Schedule: Days 1, 2, 3 and 4 of Cycles 1, 2 and 3 (every 21 days) + 2 days)
  Other Names: Cabazitaxel-PF Induction Chemotherapy
  Arms: Cabazitaxel 15mg/m2
Drug: Cabazitaxel 17.5mg/m2 — * Cabazitaxel on D1 Dose: 17.5mg/m2 IV x 1 Route: Intravenous infusion over 60 minutes, mixed as described in protocol over 1 hour Schedule: Day 1, every 21 days (+ 2 days)
  * Cisplatin on D1 Dose: 100 mg/m2 Route: Intravenous infusion over 60 minutes to 3 hours, mixed in 1000 ml of normal saline Schedule: Day 1, every 21 days (+ 2 days)
  * 5 Fluorouracil on D1-D4 Dose: 800 mg/m2/day Route: 24-hour continuous infusion over 4 days Schedule: Days 1, 2, 3 and 4 of Cycles 1, 2 and 3 (every 21 days) + 2 days)
  Other Names: Cabazitaxel-PF Induction Chemotherapy
  Arms: Cabazitaxel 17.5mg/m2
Drug: Cabazitaxel 20mg/m2 — * Cabazitaxel on D1 Dose: 20mg/m2 IV x 1 Route: Intravenous infusion over 60 minutes, mixed as described in protocol over 1 hour Schedule: Day 1, every 21 days (+ 2 days)
  * Cisplatin on D1 Dose: 100 mg/m2 Route: Intravenous infusion over 60 minutes to 3 hours, mixed in 1000 ml of normal saline Schedule: Day 1, every 21 days (+ 2 days)
  * 5 Fluorouracil on D1-D4 Dose: 800 mg/m2/day Route: 24-hour continuous infusion over 4 days Schedule: Days 1, 2, 3 and 4 of Cycles 1, 2 and 3 (every 21 days) + 2 days)
  Other Names: Cabazitaxel-PF Induction Chemotherapy
  Arms: Cabazitaxel 20mg/m2

SUMMARY:
The primary objective of this study is to determine the first-cycle maximum tolerated dose (MTD) and recommended Phase II (RP2D) dose of Cabazitaxel when combined with Cisplatin and Follow-Up induction chemotherapy in patients with locally advanced squamous cell carcinoma of the head and neck for three cycles.

DETAILED DESCRIPTION:
The primary study objectives are the following:

* To assess the safety, the maximum tolerated dose (MTD) and the dose limiting toxicity of cabazitaxel when combined with cisplatin and Follow-Up (FU) induction chemotherapy in patients with locally advanced squamous cell carcinoma of the head and neck (SCCHN).
* To establish the phase II recommended dose of cabazitaxel when combined with cisplatin and Follow-Up induction in patients with locally advanced squamous cell carcinoma of the head and neck.

The secondary study objectives, in regards to the combined Cabazitaxel-Platinum Fluorouracil regimen in patients with newly diagnosed squamous cell carcinoma of the head and neck, are the following:

* To assess the toxicity profile
* To assess best Overall Response Rate (complete and partial responses) after completion of 3 cycles of treatment
* To assess Progression Free Survival (PFS) and Overall Survival (OS) after 3 years Analysis of the secondary variables will be primarily descriptive in nature due to the small sample size. All results will be considered hypothesis generating to be confirmed in a future study.

Patient, for whom an informed consent has been obtained and who have met the inclusion/exclusion criteria after having the screening evaluation performed within a one-week window, will be assigned to a dose level according to the dose escalation rule described in the protocol. Treatment consists of an Induction chemotherapy period, which is the period when the patient will undergo 3 cycles of Cabazitaxel-Platinum Fluorouracil (PF). The Induction chemotherapy will be followed by Consolidation Therapy, which is 6-7 weeks of Chemoradiation treatment or Surgery + Recovery time, depending on their primary site and overall medical condition. Both treatment periods will consist of approximately 16 weeks (9 weeks of Induction and 7 weeks of Consolidation, if Chemoradiation Radiation Therapy (CRT)), or shorter than 16 weeks, if surgery. After three cycles, the patients will be assessed for clinical, radiographic, and pathologic response to Cabazitaxel-Platinum Fluorouracil before beginning Chemoradiation Radiation Therapy or surgery. Patients, who do not complete three cycles of Cabazitaxel-Platinum Fluorouracil for reasons of toxicity, progressive disease, choice, or other medical necessity, will be treated with standard Chemoradiation Radiation Therapy or surgery depending on their primary site and overall medical condition. Once the Consolidation treatment is completed, the follow-up of patients will be for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage IV only, previously untreated, locally advanced SCCHN (patients may have had previous surgery, but not chemotherapy or radiotherapy).
* During the dose escalation phase before the MTD and DLT are established for cabazitaxel combined with cisplatin and FU induction chemotherapy primary sites allowed include the oral cavity, oropharynx, larynx, hypopharynx, nasopharynx, and unknown primary regardless of Human Papilloma Virus (HPV) status. Metastatic SCCHN will be allowed in escalation phase.
* Once MTD and DLT for cabazitaxel combined with cisplatin and FU induction chemotherapy are established (expansion cohort) primary sites allowed include the oral cavity, oropharynx (HPV negative only), larynx, hypopharynx, nasopharynx, and unknown primary (HPV negative only). No patients with metastases will be allowed in this phase (expansion cohort).
* Age >/= 18 years
* Eastern Cooperative Oncology Group PS 0-1
* Predicted life expectancy >/= 12 weeks
* Absolute Neutrophilic Count (ANC) >/= 1.5 x 10^9/L, Platelets >/= 100 x 10^9/L; bilirubin </= 1.5 x Upper Limit of Normal (ULN), Aspartate Aminotransferase (AST) and/or Alanine Aminotransferase (ALT) </= 2.5 x ULN or </= 5 x ULN if patient has documented liver metastases; serum creatinine </= 1.5 x ULN
* Patients in the expansion cohorts must have measurable disease per Response Evaluation Criteria in Solid Tumors(RECIST)
* Patients must be accessible for repeat dosing and follow-up
* Patients - both males and females - with reproductive potential must agree to practice effective contraceptive measures throughout the study. Women of childbearing potential must provide a negative pregnancy test at baseline and on Day 1
* Patients must provide verbal and written informed consent to participate in the study

Exclusion Criteria:

* Locally advanced HPV positive oropharyngeal or unknown primary SCCHN for the expansion cohort only (Once MTD and DLT for cabazitaxel combined with cisplatin and FU induction chemotherapy established).
* History of significant cardiac disease unless the disease is well-controlled
* Grade 2 peripheral neuropathy
* No excessive alcohol consumption will be allowed
* Serious comorbid illness, and involuntary weight loss of more than 20% of body weight in the 3 months preceding study entry
* History of cerebrovascular accident (CVA) within 12 months prior to registration or that is not stable
* History of any psychiatric condition that might impair the patient's ability to understand or to comply with the requirements of the study or to provide informed consent
* Pregnant or breast-feeding females Gastrointestinal (GI) abnormalities including inability to take oral medication, requirement for IV alimentation, active peptic ulcer, or prior surgical procedures affecting absorption
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the study drug
* Any type of active seizure disorder
* Use of drugs that have a risk of causing QT interval prolongation within 14 days prior to Day 1 dosing
* Use of strong or moderate CYP3A4 or CYP1A2 inhibitors/inducers, with the exception of low-dose steroids, within 14 days prior to Day 1 dosing
* Symptomatic brain metastases that are not stable, require steroids, or that have required radiation within the last 28 days
* Active or uncontrolled infections or serious illnesses or medical conditions that could interfere with the patient's ongoing participation in the study
* History of Hepatitis C or Human Immunodeficiency Virus (HIV) infection, autoimmune disease, or major organ transplant.
* Surgery, irradiation or chemotherapy within the previous 4 weeks
* Any other concomitant anticancer therapies
* Patients will be excluded if they received any prior chemotherapy, radiotherapy, or treatment with biologic response modifiers (except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix)
* History of colitis or chronic diarrheal illness
* History of, or active, co-morbid medical condition, which in the opinion of the investigator, would raise significant risk to the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | at 1 week
  MTD is defined as the dose level immediately below the DLT. The study will be conducted until MTD and recommended Phase II dose are established.
Maximum Tolerated Dose (MTD) | at 4 weeks
  MTD is defined as the dose level immediately below the DLT. The study will be conducted until MTD and recommended Phase II dose are established.
Maximum Tolerated Dose (MTD) | at 7 weeks
  MTD is defined as the dose level immediately below the DLT. The study will be conducted until MTD and recommended Phase II dose are established.
Maximum Tolerated Dose (MTD) | at 9 weeks
  MTD is defined as the dose level immediately below the DLT. The study will be conducted until MTD and recommended Phase II dose are established.
Dose-limiting toxicity (DLT) | at 1 week
  DLT is defined as a grade3 toxicity lasting more than 7 days or grade 4 or 5 toxicity, with the exception of febrile neutropenia which will be considered as ½ DLT per full dose per episode. The DLT will be the basis for determining the MTD. Treatment cohorts will be dosed in escalating order only after the safety of the previous dose level is established, or until an MTD has been determined.
Dose-limiting toxicity (DLT) | at 4 weeks
  DLT is defined as a grade3 toxicity lasting more than 7 days or grade 4 or 5 toxicity, with the exception of febrile neutropenia which will be considered as ½ DLT per full dose per episode. The DLT will be the basis for determining the MTD. Treatment cohorts will be dosed in escalating order only after the safety of the previous dose level is established, or until an MTD has been determined.
Dose-limiting toxicity (DLT) | at 7 weeks
  DLT is defined as a grade3 toxicity lasting more than 7 days or grade 4 or 5 toxicity, with the exception of febrile neutropenia which will be considered as ½ DLT per full dose per episode. The DLT will be the basis for determining the MTD. Treatment cohorts will be dosed in escalating order only after the safety of the previous dose level is established, or until an MTD has been determined.
Dose-limiting toxicity (DLT) | at 9 weeks
  DLT is defined as a grade3 toxicity lasting more than 7 days or grade 4 or 5 toxicity, with the exception of febrile neutropenia which will be considered as ½ DLT per full dose per episode. The DLT will be the basis for determining the MTD. Treatment cohorts will be dosed in escalating order only after the safety of the previous dose level is established, or until an MTD has been determined.

SECONDARY OUTCOMES:
Toxicity Profile | at 9 weeks
  The toxicity profile of cabazitaxel when combined with cisplatin and FU induction chemotherapy will be assessed
Overall Response Rate | at 9 weeks
  The Best Overall Response Rate (complete and partial responses) will be assessed after completion of 3 cycles of treatment.
Progression Free Survival/Overall Survival | for 3 years
  The Progression Free Survival and Overall Survival will be assessed during the 3-year follow-up period. The follow-up period is every 3 months for the first 2 years post consolidation (week 16) thereafter every 6 months for the 3rd year post consolidation (week 16).

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Misiukiewicz, M.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Forastiere AA, Goepfert H, Maor M, Pajak TF, Weber R, Morrison W, Glisson B, Trotti A, Ridge JA, Chao C, Peters G, Lee DJ, Leaf A, Ensley J, Cooper J. Concurrent chemotherapy and radiotherapy for organ preservation in advanced laryngeal cancer. N Engl J Med. 2003 Nov 27;349(22):2091-8. doi: 10.1056/NEJMoa031317. PMID 14645636
- [Background] Adelstein DJ, Li Y, Adams GL, Wagner H Jr, Kish JA, Ensley JF, Schuller DE, Forastiere AA. An intergroup phase III comparison of standard radiation therapy and two schedules of concurrent chemoradiotherapy in patients with unresectable squamous cell head and neck cancer. J Clin Oncol. 2003 Jan 1;21(1):92-8. doi: 10.1200/JCO.2003.01.008. PMID 12506176
- [Background] Domenge C, Hill C, Lefebvre JL, De Raucourt D, Rhein B, Wibault P, Marandas P, Coche-Dequeant B, Stromboni-Luboinski M, Sancho-Garnier H, Luboinski B; French Groupe d'Etude des Tumeurs de la Tete et du Cou (GETTEC). Randomized trial of neoadjuvant chemotherapy in oropharyngeal carcinoma. French Groupe d'Etude des Tumeurs de la Tete et du Cou (GETTEC). Br J Cancer. 2000 Dec;83(12):1594-8. doi: 10.1054/bjoc.2000.1512. PMID 11189100
- [Background] Posner MR, Hershock DM, Blajman CR, Mickiewicz E, Winquist E, Gorbounova V, Tjulandin S, Shin DM, Cullen K, Ervin TJ, Murphy BA, Raez LE, Cohen RB, Spaulding M, Tishler RB, Roth B, Viroglio Rdel C, Venkatesan V, Romanov I, Agarwala S, Harter KW, Dugan M, Cmelak A, Markoe AM, Read PW, Steinbrenner L, Colevas AD, Norris CM Jr, Haddad RI; TAX 324 Study Group. Cisplatin and fluorouracil alone or with docetaxel in head and neck cancer. N Engl J Med. 2007 Oct 25;357(17):1705-15. doi: 10.1056/NEJMoa070956. PMID 17960013
- [Background] Jordan MA, Wilson L. Microtubules as a target for anticancer drugs. Nat Rev Cancer. 2004 Apr;4(4):253-65. doi: 10.1038/nrc1317. No abstract available. PMID 15057285
- [Background] Mita AC, Denis LJ, Rowinsky EK, Debono JS, Goetz AD, Ochoa L, Forouzesh B, Beeram M, Patnaik A, Molpus K, Semiond D, Besenval M, Tolcher AW. Phase I and pharmacokinetic study of XRP6258 (RPR 116258A), a novel taxane, administered as a 1-hour infusion every 3 weeks in patients with advanced solid tumors. Clin Cancer Res. 2009 Jan 15;15(2):723-30. doi: 10.1158/1078-0432.CCR-08-0596. PMID 19147780
- [Background] de Bono JS, Oudard S, Ozguroglu M, Hansen S, Machiels JP, Kocak I, Gravis G, Bodrogi I, Mackenzie MJ, Shen L, Roessner M, Gupta S, Sartor AO; TROPIC Investigators. Prednisone plus cabazitaxel or mitoxantrone for metastatic castration-resistant prostate cancer progressing after docetaxel treatment: a randomised open-label trial. Lancet. 2010 Oct 2;376(9747):1147-54. doi: 10.1016/S0140-6736(10)61389-X. PMID 20888992
- [Background] Rooney M, Kish J, Jacobs J, Kinzie J, Weaver A, Crissman J, Al-Sarraf M. Improved complete response rate and survival in advanced head and neck cancer after three-course induction therapy with 120-hour 5-FU infusion and cisplatin. Cancer. 1985 Mar 1;55(5):1123-8. doi: 10.1002/1097-0142(19850301)55:53.0.co;2-8. PMID 4038469
- [Background] Kish J, Drelichman A, Jacobs J, Hoschner J, Kinzie J, Loh J, Weaver A, Al-Sarraf M. Clinical trial of cisplatin and 5-FU infusion as initial treatment for advanced squamous cell carcinoma of the head and neck. Cancer Treat Rep. 1982 Mar;66(3):471-4. PMID 7037180
- [Background] Gillison ML, Koch WM, Capone RB, Spafford M, Westra WH, Wu L, Zahurak ML, Daniel RW, Viglione M, Symer DE, Shah KV, Sidransky D. Evidence for a causal association between human papillomavirus and a subset of head and neck cancers. J Natl Cancer Inst. 2000 May 3;92(9):709-20. doi: 10.1093/jnci/92.9.709. PMID 10793107
- [Background] Martinez I, Wang J, Hobson KF, Ferris RL, Khan SA. Identification of differentially expressed genes in HPV-positive and HPV-negative oropharyngeal squamous cell carcinomas. Eur J Cancer. 2007 Jan;43(2):415-32. doi: 10.1016/j.ejca.2006.09.001. Epub 2006 Oct 31. PMID 17079134
- [Background] Cullen KJ, Schumaker L, Nikitakis N, Goloubeva O, Tan M, Sarlis NJ, Haddad RI, Posner MR. beta-Tubulin-II expression strongly predicts outcome in patients receiving induction chemotherapy for locally advanced squamous carcinoma of the head and neck: a companion analysis of the TAX 324 trial. J Clin Oncol. 2009 Dec 20;27(36):6222-8. doi: 10.1200/JCO.2009.23.0953. Epub 2009 Nov 16. PMID 19917838
- [Background] Shiga H, Heath EI, Rasmussen AA, Trock B, Johnston PG, Forastiere AA, Langmacher M, Baylor A, Lee M, Cullen KJ. Prognostic value of p53, glutathione S-transferase pi, and thymidylate synthase for neoadjuvant cisplatin-based chemotherapy in head and neck cancer. Clin Cancer Res. 1999 Dec;5(12):4097-104. PMID 10632346
- [Background] Nishimura T, Shiga H, Wakisaka N, Furukawa M. [Glutathione and cisplatin resistance in head and neck cancer]. Nihon Jibiinkoka Gakkai Kaiho. 1999 Feb;102(2):236-42. doi: 10.3950/jibiinkoka.102.236. Japanese. PMID 10191625
- [Background] Cullen KJ, Newkirk KA, Schumaker LM, Aldosari N, Rone JD, Haddad BR. Glutathione S-transferase pi amplification is associated with cisplatin resistance in head and neck squamous cell carcinoma cell lines and primary tumors. Cancer Res. 2003 Dec 1;63(23):8097-102. PMID 14678959
- [Background] Forastiere A, Koch W, Trotti A, Sidransky D. Head and neck cancer. N Engl J Med. 2001 Dec 27;345(26):1890-900. doi: 10.1056/NEJMra001375. No abstract available. PMID 11756581
- [Background] Temam S, Flahault A, Perie S, Monceaux G, Coulet F, Callard P, Bernaudin JF, St Guily JL, Fouret P. p53 gene status as a predictor of tumor response to induction chemotherapy of patients with locoregionally advanced squamous cell carcinomas of the head and neck. J Clin Oncol. 2000 Jan;18(2):385-94. doi: 10.1200/JCO.2000.18.2.385. PMID 10637254
- [Background] Cabelguenne A, Blons H, de Waziers I, Carnot F, Houllier AM, Soussi T, Brasnu D, Beaune P, Laccourreye O, Laurent-Puig P. p53 alterations predict tumor response to neoadjuvant chemotherapy in head and neck squamous cell carcinoma: a prospective series. J Clin Oncol. 2000 Apr;18(7):1465-73. doi: 10.1200/JCO.2000.18.7.1465. PMID 10735894
- [Background] Perrone F, Bossi P, Cortelazzi B, Locati L, Quattrone P, Pierotti MA, Pilotti S, Licitra L. TP53 mutations and pathologic complete response to neoadjuvant cisplatin and fluorouracil chemotherapy in resected oral cavity squamous cell carcinoma. J Clin Oncol. 2010 Feb 10;28(5):761-6. doi: 10.1200/JCO.2009.22.4170. Epub 2010 Jan 4. PMID 20048189
- [Background] Alsner J, Sorensen SB, Overgaard J. TP53 mutation is related to poor prognosis after radiotherapy, but not surgery, in squamous cell carcinoma of the head and neck. Radiother Oncol. 2001 May;59(2):179-85. doi: 10.1016/s0167-8140(01)00301-2. PMID 11325447
- [Background] Pena JC, Thompson CB, Recant W, Vokes EE, Rudin CM. Bcl-xL and Bcl-2 expression in squamous cell carcinoma of the head and neck. Cancer. 1999 Jan 1;85(1):164-70. doi: 10.1002/(sici)1097-0142(19990101)85:13.0.co;2-q. PMID 9921989
- [Background] Rischin D, Young RJ, Fisher R, Fox SB, Le QT, Peters LJ, Solomon B, Choi J, O'Sullivan B, Kenny LM, McArthur GA. Prognostic significance of p16INK4A and human papillomavirus in patients with oropharyngeal cancer treated on TROG 02.02 phase III trial. J Clin Oncol. 2010 Sep 20;28(27):4142-8. doi: 10.1200/JCO.2010.29.2904. Epub 2010 Aug 9. PMID 20697079
- [Background] Ang KK, Harris J, Wheeler R, Weber R, Rosenthal DI, Nguyen-Tan PF, Westra WH, Chung CH, Jordan RC, Lu C, Kim H, Axelrod R, Silverman CC, Redmond KP, Gillison ML. Human papillomavirus and survival of patients with oropharyngeal cancer. N Engl J Med. 2010 Jul 1;363(1):24-35. doi: 10.1056/NEJMoa0912217. Epub 2010 Jun 7. PMID 20530316
- [Background] Paccagnella A, Ghi MG, Loreggian L, Buffoli A, Koussis H, Mione CA, Bonetti A, Campostrini F, Gardani G, Ardizzoia A, Dondi D, Guaraldi M, Cavallo R, Tomio L, Gava A; Gruppo di Studio Tumori della Testa e del Collo XRP 6976 F/2501 Study. Concomitant chemoradiotherapy versus induction docetaxel, cisplatin and 5 fluorouracil (TPF) followed by concomitant chemoradiotherapy in locally advanced head and neck cancer: a phase II randomized study. Ann Oncol. 2010 Jul;21(7):1515-1522. doi: 10.1093/annonc/mdp573. Epub 2009 Dec 23. PMID 20032123
- [Background] Pivot X, Koralewski P, Hidalgo JL, Chan A, Goncalves A, Schwartsmann G, Assadourian S, Lotz JP. A multicenter phase II study of XRP6258 administered as a 1-h i.v. infusion every 3 weeks in taxane-resistant metastatic breast cancer patients. Ann Oncol. 2008 Sep;19(9):1547-52. doi: 10.1093/annonc/mdn171. Epub 2008 Apr 23. PMID 18436520
- [Background] El-Mofty SK, Patil S. Human papillomavirus (HPV)-related oropharyngeal nonkeratinizing squamous cell carcinoma: characterization of a distinct phenotype. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):339-45. doi: 10.1016/j.tripleo.2005.08.001. PMID 16504868